CLINICAL TRIAL: NCT01282073
Title: A Randomized Controlled Multi-center Trial of Mycophenolate Mofetil for the Patient With High Risk Membranous Nephropathy
Brief Title: Mycophenolate Mofetil in Patients With Progressive Idiopathic Membranous Nephropathy
Acronym: MMFPRIMER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyungpook National University Hospital (Other)
Collaborators: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Principal Investigator, Sun-Hee Park, Professor, Kyungpook National University Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MMFPRIMER
Record Dates: First submitted 2011-01-19; First posted 2011-01-24 (Estimated); Results first posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Glomerulonephritis, Membranous
Keywords: Idiopathic membranous nephropathy; Mycophenolate mofetil; Proteinuria; Renal function
MeSH Terms: conditions — Glomerulonephritis, Membranous; Proteinuria | interventions — Mycophenolic Acid; Steroids; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mycophenolate mofetil, low dose steroid (Experimental)
  Interventions: Drug: Mycophenolate mofetil, low dose steroid
- Cyclosporin, low dose steroid (Active Comparator)
  Interventions: Drug: Cyclosporin, low dose steroid

INTERVENTIONS:
Drug: Mycophenolate mofetil, low dose steroid — Mycophenolate Mofetil: Myconol capsule 250mg, Myconol 500 mg bid per day (less than 50kg), 750 ~ 1000 mg bid per day (more than 50kg)
  Steroid: Methylprednisone 4mg tablet or Prednisolone 5mg tablet or Deflazacort 6mg tablet. Prednisolone dose: 0.15mg/kg up to a maximum dose of 15mg/day
  Duration: 48 weeks
  Other Names: Myconol, MMF
  Arms: Mycophenolate mofetil, low dose steroid
Drug: Cyclosporin, low dose steroid — Cyclosporin: Implanta soft cap (cyclosporin microemulsion) 25mg/100mg, starting dose of 4mg/kg per day and titrate according to investigator's decision based on cyclosporin trough level (100±50 ng/ml)
  Steroid: same dosage with active comparator goup
  Duration: 48 weeks
  Other Names: Implanta soft capsule
  Arms: Cyclosporin, low dose steroid

SUMMARY:
Cyclosporin decreases proteinuria and improve renal function in patients with idiopathic membranous nephropathy, but has a risk of side effects such as nephrotoxicity. The investigators plan to the study to evaluate whether mycophenolate mofetil (MMF) could be a reasonable alternative with fewer side effect.

DETAILED DESCRIPTION:
Idiopathic membranous nephropathy is most common cause of glomerulonephritis in adults. Persistent high grade proteinuria or progressively decrease of renal function is a risk factor for end stage renal disease in idiopathic membranous nephropathy. It has been reported that cyclosporin in patients with idiopathic membranous nephropathy decreases proteinuria and improve renal function. Mycophenolate mofetil is a recently developed immunosuppressive agent with fewer side effect than cyclosporin. In this study patients with high risk group of progressive idiopathic membranous nephropathy will be treated with mycophenolate mofetil and low dose prednisone. The outcome will be compared to controls treated with cyclosporin and low dose prednisone.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with idiopathic membranous nephropathy
2. The duration of disease is less than twelve months
3. Patients with persistent proteinuria more than 8 grams per day
4. Patients who provided informed consent
5. The cases that satisfy more than three of following items even if proteinuria is less than 8 grams per day:

   * eGFR < 60 ml/min/1.73m2
   * Hypertension (BP above 140/90mmHg or BP above 120/80 in patients taking anti-hypertensive agents)
   * 24 hours urine protein or spot urine protein/creatinine ratio > 5.0 g/day
   * Serum albumin (g/dL) < 3.0
   * Selectivity index > 0.2

Exclusion Criteria:

1. Severe digestive organ disease
2. Allergy history to clinical trial medication and acute or chronic allergy for 4 weeks recently.
3. Clinical history of treatment with other immunosuppressive medication
4. Probability of pregnancy, breast feeding woman
5. Uncontrolled hypertension (more than 160/100mmHg)
6. Uncontrolled systemic disease
7. Drug addiction or alcoholics within 6 months
8. eGFR is less than 30ml/min at screening
9. Abnormal liver function test (more than 3 times above compared with normal value)
10. Absolute neutrophil count <1,500/mm3 or leukocyte <2,500/mm3 or platelets <100,000/mm3
11. Secondary membranous nephropathy
12. Expected life expectancy is less than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sun-Hee Park, MD, Principal Investigator — Kyungpook National University Hospital
Locations (9):
- South Korea (9):
  - Dong-A University Medical Center, Busan
  - Inje University Haeundae Paik Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Daegu Fatima Hospital, Daegu
  - Yeungnam University Medical Center, Daegu
  - Seoul National University Hospital, Seoul
  - Yonsei University Hospital, Seoul
  - Boramae Medical Center, Seoul
  - Ulsan University Hospital, Ulsan

REFERENCES:
- [Derived] von Groote TC, Williams G, Au EH, Chen Y, Mathew AT, Hodson EM, Tunnicliffe DJ. Immunosuppressive treatment for primary membranous nephropathy in adults with nephrotic syndrome. Cochrane Database Syst Rev. 2021 Nov 15;11(11):CD004293. doi: 10.1002/14651858.CD004293.pub4. PMID 34778952
- [Derived] Choi JY, Kim DK, Kim YW, Yoo TH, Lee JP, Chung HC, Cho KH, An WS, Lee DH, Jung HY, Cho JH, Kim CD, Kim YL, Park SH. The Effect of Mycophenolate Mofetil versus Cyclosporine as Combination Therapy with Low Dose Corticosteroids in High-risk Patients with Idiopathic Membranous Nephropathy: a Multicenter Randomized Trial. J Korean Med Sci. 2018 Feb 26;33(9):e74. doi: 10.3346/jkms.2018.33.e74. PMID 29441742

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mycophenolate Mofetil, Low Dose Steroid | Cyclosporin, Low Dose Steroid
Started | 21 | 18
Completed | 21 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mycophenolate Mofetil, Low Dose Steroid | Cyclosporin, Low Dose Steroid | Total
Number analyzed (Participants) | 21 | 18 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (10.0) | 52.7 (10.9) | 55.4 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 16 | 9 | 25
Region of Enrollment [Number; unit: participants]
  South Korea | 21 | 18 | 39

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Complete Remission
Description: Complete remission: Reduction in proteinuria to 200 mg per day with stable serum albumin with more than 3.5 g/dL
Time Frame: at 48 week after treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Mycophenolate Mofetil, Low Dose Steroid | Cyclosporin, Low Dose Steroid
Number analyzed (Participants) | 21 | 18
Participants | 4 | 3

2. Primary Outcome: Percentage of Partial Remission
Description: Partial remission: Reduction in proteinuria to greater than 50 percent of initial values or absolute values of proteinuria between 200 mg and 3.5 g per day
Time Frame: at 48 week after treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Mycophenolate Mofetil, Low Dose Steroid | Cyclosporin, Low Dose Steroid
Number analyzed (Participants) | 21 | 18
Participants | 12 | 9

3. Secondary Outcome: Estimated Glomerular Filtration Rate (eGFR)
Description: The change of eGFR mesured by Modification of Diet in Renal Disease (MDRD) study equation from baseline to 1 year after treatment
Time Frame: at 48 week after treatment
Reporting Status: Not Posted

4. Secondary Outcome: Relapse
Description: A relapse is return of proteinuria to approximately 3.5g/day in patients who had previously undergone a complete or partial remission
Time Frame: For 48 weeks after treatment
Reporting Status: Not Posted

5. Secondary Outcome: Proteinuria
Description: The change of proteinuria from baseline to 48 week after treatment
Time Frame: at 48 week after treatment
Reporting Status: Not Posted

6. Secondary Outcome: Side Effects
Description: Any undesired effects of interventional drugs
Time Frame: For 48 weeks after treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 48 weeks
Arm/Group | Mycophenolate Mofetil, Low Dose Steroid | Cyclosporin, Low Dose Steroid
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/18
Other Adverse Events (participants affected / at risk) | 12/21 | 9/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mycophenolate Mofetil, Low Dose Steroid (N=21) | Cyclosporin, Low Dose Steroid (N=18)
Diarrhea (Gastrointestinal disorders) | 2 | 2
Epigastric discomfort (Gastrointestinal disorders) | 3 | 4
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Upper respiratory infection (Infections and infestations) | 6 | 3
Urinary tract infection (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 2 | 1
New onset diabetes mellitus (Endocrine disorders) | 1 | 1
Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No